CLINICAL TRIAL: NCT06393049
Title: Microdialysis and Jugular Bulb Glucose Profiles During Hyperglycaemic Clamping in Patients with Severe Acute Brain Injury
Acronym: CLAMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne-Sophie Worm Fenger, Principal investigator, MD, PhD fellow, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23072860
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Acute Brain Injury
Keywords: Acute brain injury; Intensive care; Neurointensive care; Anaesthesiology; Multimodal neuromonitoring; Glucose; Hyperglycaemic clamp
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: 14 patients, all will have an hyperglycaemic clamp performed during admission while measuring cerebral microdialysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperglycaemic clamp (Other): The purpose of hyperglycaemic clamping is to raise the blood glucose level to a fixed plateau and maintain the plateau for at least one hour to observe a steady-state blood glucose concentration.
  The investigators intend to perform the hyperglycaemic clamping procedure one time in all 14 patients following an overnight fast and aim for a fixed blood glucose level above 8 mmol/L.
  The patient will have an arterial line placed in the radial artery, a retrograde catheterization of the jugular bulb and a venous line for infusions of glucose, potassium, and isotonic saline.
  To maintain potassium levels at wanted levels, an isotonic saline solution containing potassium will be infused continuously and arterial samples of potassium and glucose will be measured at minimum every 10 minutes from the start of the intervention.
  Interventions: Other: Hyperglycaemic clamp

INTERVENTIONS:
Other: Hyperglycaemic clamp — Following an overnight fast, the investigators will perform simultaneous samples from the arterial line, the venous line, and microdialysis and consider these samples as baseline values.
  If the patient's blood glucose level is at 8-10 mmol/L at baseline, the investigators will not proceed with the intervention and instead evaluate if the intervention can take place the following day.
  After baseline values are measured, intravenous glucose 20% (200g/1,000 ml) is infused to raise the glucose levels in both plasma and extravascular glucose compartments with approximately 3 mmol/L.

SUMMARY:
Acute brain injury is a serious condition that often results in admission to an intensive care unit. Some of the most seriously ill patients are fitted with multimodal neuromonitoring, a newer monitoring modality that can, among other things, measure oxygen tension and sugar levels in brain tissue. It is common clinical practice, but the interaction between the body's sugar levels and the brain's sugar levels is not sufficiently elucidated.

The study will investigate the relationship between the body's sugar levels, measured in arterial and venous blood, and the brain's sugar level, measured by microdialysis, in patients with severe acute brain injury.

Furthermore, we hope to be able to use our measurements to set up a mathematical model for the brain's sugar uptake.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Admission to the neuro-ICU at Rigshospitalet.
* Multimodal neuromonitoring

Exclusion Criteria:

* Closest relative does not understand written and spoken Danish or English.
* Patients with known diabetes mellitus upon admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
(Change in) MD-glucose (mmol/L) | Throughout the intervention, approximately five hours
  Change in) MD-glucose (mmol/L) over time as a function of (a set change in) arterial blood glucose (mmol/L)

SECONDARY OUTCOMES:
Jugular vein glucose (mmol/L) over time as a function of arterial blood glucose. | Throughout the intervention, approximately five hours
  Jugular vein glucose (mmol/L) over time as a function of arterial blood glucose (mmol/L)
Lactate-pyruvate-ratio (LP-ratio) as a function of arterial blood glucose. | Throughout the intervention, approximately five hours.
  Two other microdialysis paramethers, lactate and pyruvat, will be assessed to evaluate the lactate-pyruvate ratio over time as a function of arteriel blood glucose.

OTHER OUTCOMES:
Mathematic model of transport of glucose over the blood brain barrier. | Throughout the intervention, approximately five hours.
  Mathematic model of transport of glucose over the blood brain barrier.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Neuroanaesthesiology, Rigshospitalet, Copenhagen
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No